CLINICAL TRIAL: NCT02850523
Title: Cognitive Behavioural Group Therapy for Perinatal Anxiety: A Randomized Controlled Trial
Brief Title: Cognitive Behavioural Group Therapy for Perinatal Anxiety
Acronym: CBT-PA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Sheryl Green, Cinical Health Psychologist, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCRA-SG2
Record Dates: First submitted 2016-07-26; First posted 2016-08-01 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Perinatal Anxiety
Keywords: Cognitive-behavioural therapy (CBT)
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: A single-blind, randomized controlled trial was conducted to evaluate the effectiveness of a new group-based cognitive-behavioural therapy (CBGT) for women with anxiety during pregnancy or in the early postpartum.
Who Masked: Outcomes Assessor
Masking Description: Assessors conducted assessments of symptoms and overall functioning at baseline, 6-weeks post-baseline, and (for participants assigned to CBGT) at 3-months post-treatment. Assessors were unaware of participants' assigned condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): After an initial assessment, the experimental group will receive 6 weekly sessions (2 hours long) of group Cognitive Behavioural Therapy for Perinatal Anxiety (n=6 per group) for perinatal anxiety. They will then be re-assessed at post-treatment and 3 months post-treatment to determine the effectiveness of the treatment and whether these effects are maintained 3 months after treatment.
  Interventions: Other: Cognitive Behavioural Therapy for Perinatal Anxiety
- Waitlist Control (No Intervention): After an initial assessment, the wait-list control group will not receive any treatment for 6 weeks. They will then be re-assessed after 6 weeks and this data will be used to compare this group to the experimental group to determine the effectiveness of the treatment. After this re-assessment they will be offered the same treatment as the experimental group: 6 weekly sessions (2 hours long) of group Cognitive Behavioural Therapy for Perinatal Anxiety

INTERVENTIONS:
Other: Cognitive Behavioural Therapy for Perinatal Anxiety — The treatment consists of cognitive and behavioural strategies for treating anxiety, tailored specifically to a perinatal/postpartum population.
  Arms: Experimental

SUMMARY:
This study evaluated the effectiveness of a 6-week, group-based, cognitive behavioural therapy (CGBT) program for women with anxiety disorders (with or without comorbid depressive symptoms) during pregnancy or early postpartum. The CBGT program was evaluated compared to a 6-week waitlist condition.

DETAILED DESCRIPTION:
Anxiety disorders affect up to 15% of women in the perinatal period (i.e., pregnancy, postpartum) and are a serious mental health concern. Anxiety disorders often coexist with depression and result in high distress and an impaired ability for new mothers to take care of themselves and their babies. In spite of the high prevalence of anxiety disorders during pregnancy and postpartum, research and clinical attention in this area is lacking and no empirically supported psychological treatments exist. Further, since many pregnant or postpartum women are unable or choose not to take medication for their mental health symptoms, establishing an effective non-pharmacological alternative is imperative. Cognitive-behavioural therapy is a well established psychological treatment for anxiety and mood disorders, with moderate to large effect sizes (Cohen's d = 0.5-1.3). The investigators developed a novel group-based cognitive-behavioural treatment program (CBGT) for perinatal women with anxiety disorders. In an initial, single-sample pilot study (Green et al., 2015), a significant reduction in symptoms of anxiety and depression was found from pre to post-treatment, along with reported high levels of treatment satisfaction. The purpose of the current study is to evaluate the effectiveness of this treatment using a larger sample and a randomized controlled trial (RCT).

ELIGIBILITY:
Eligibility criteria:

1. 18-45 years of age
2. pregnant or within the first six months postpartum
3. principal diagnosis of an anxiety disorder with or without comorbid depression
4. not taking psychoactive medication or, if taking these medications, no change in dose and type ≥ 6 weeks prior to the baseline assessment
5. no changes in psychoactive medication during the 6-week CBT treatment or 6-week waitlist
6. fluent in English

Exclusion criteria:

1. severe depression or active suicidal ideation
2. current psychosis or substance use disorder

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
State-Trait Inventory of Cognitive and Somatic Anxiety (STICSA) | 6 weeks
  Changes in anxiety symptoms will be assessed through the State-Trait Inventory for Cognitive and Somatic Anxiety (STICSA; Gros et al.,2007) to examine whether CBT for perinatal anxiety is effective in reducing anxiety symptoms. Items on the STICSA are rated on a 4-point likert scale ranging from 1 (not at all) to 4 (very much so), with higher scores indicating worse anxiety symptoms. The STICSA has two subscales (i.e., cognitive subscale and somatic subscale) and a total score that will be used in analysis. Ten items comprise the cognitive subscale, meaning scores can range from 10-40. Eleven items comprise the somatic subscale, meaning scores can range from 11 -44. The total score is a sum of both subscales with possible total scores in the range of 21-84.

SECONDARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) | 6 weeks
  Changes in mood symptoms will be assessed through the Edinburgh Postnatal Depression Scale (EPDS; Cox et al., 1987) to examine whether CBT for perinatal anxiety is effective in reducing mood symptoms. Items on the EPDS are rated from 0-3, with higher total scores indicating more depressive symptoms. Possible scores on the EPDS range from 0-30. A clinical cut-off of 13 is used to indicate probable depression.
Penn State Worry Questionnaire (PSWQ) | 6 weeks
  Changes in worry symptoms will be assessed through the Penn State Worry Questionnaire (PSWQ; Meyer et al.,1990) to examine whether CBT for perinatal anxiety is effective in reducing worry. Items on the PSWQ are rated from 1 (not at all typical of me) to 5 (very typical of me), with higher total scores indicating higher levels of worry. Scores on the PSWQ can range from 16 to 80.
Intolerance of Uncertainty Scale (IUS-12) | 6 weeks
  Changes in intolerance of uncertainty will be assessed through the Intolerance of Uncertainty Scale (IUS-12; Carleton, R. N., Norton, M. P. J., & Asmundson, G. J, 2007) to examine whether CBT for perinatal anxiety is effective in reducing intolerance of uncertainty. Items on the IUS-12 are rated on a 5-point likert scale ranging from 1 (not at all characteristic of me) to 5 (entirely characteristic of me). Higher scores indicate great levels of intolerance of uncertainty and are associated with worse outcomes. The IUS-12 has a total score, along with two subscale scores. The prospective anxiety subscale comprises of seven items, with possible scores ranging from 7-35. The inhibitory anxiety scale comprises of five items, with possible scores ranging from 5-25. The total IUS-12 score is calculated by summing the two subscales, meaning total scores range from 12-60.
Multidimensional Perfectionism Scale (MPS) | 6 weeks
  Changes in general perfectionism symptoms will be assessed through the Multidimensional perfectionism scale (MPS; Hewitt et al.,1991) to examine whether CBT for perinatal anxiety is effective in reducing perfectionism. Items on the MPS are rated on a 7-point scale ranging from 1-7. The MPS is comprised of three subscales with 15 items each that measure self-oriented perfectionism, other-oriented perfectionism, and socially prescribed perfectionism. Scores on each subscale range from 15-105, with higher scores indicating greater levels of that type of perfectionism. A total score on the MPS can be obtained by summing the three subscales making the total score range 45-315.
Multidimensional Parenting Perfectionism Scale (MPPQ) | 6 weeks
  Changes in parenting perfectionism symptoms will be assessed through the Multidimensional parenting perfectionism scale (MPPQ; Snell, 1997) to examine whether CBT for perinatal anxiety is effective in reducing parental perfectionism. Items on the MPPQ are rated on a 5-point scale ranging from 0 (not at all characteristic of me) to 4 (very characteristic of me) , with higher scores indicating greater amounts of parental perfectionism. The MPPQ has 11 subscales. Each subscale has 5-items with scores ranging from 0-20. Total scores are obtained by summing all subscale scores and can range from 0-260.
Parenting Sense of Competence Scale (PSOC) | 6 weeks
  Changes in parenting competence will be assessed through Parenting Sense of Competence Scale (PSOC; Gibaud-Wallston & Wandersman, 1978) to examine whether CBT for perinatal anxiety is effective in increasing sense of competence. Items on the PSOC are rated from 1 (strongly disagree) to 6 (strongly agree), with total scores on the PSOC ranging from 17-102. Higher total scores on the PSOC indicate a higher sense of parenting competency.
Social Provisions Scale (SPS) | 6 weeks
  Social support will be assessed through the Social Provisions Scale (SPS; Cutrona & Russell, 1987) to examine whether CBT for perinatal anxiety is effective in increasing the degree to which the participant's social relationships provide dimensions of social support. Items on the SPS are rated on a 4-point scale ranging from 1-4. Total scores on the SPS range from 24-96, with higher scores indicating greater social support.
Abbreviated Dyadic Adjustment Scale (ADAS) | 6 weeks
  Changes in relationship satisfaction will be assessed through Abbreviated Dyadic Adjustment Scale (ADAS; Spanier, 1976) to examine whether CBT for perinatal anxiety is effective in increasing the self-reported quality of marital and other close relationships. Items 1-6 on the ADAS are rated on a 6-point scale ranging from 0-5. Item 7 is rated on a 7-point scale ranging from 0 (extremely unhappy) to 6 (perfect) and provides a happiness rating. Item 7 is not included in the total score for the ADAS, meaning total scores can range from 0-30. Higher scores on the ADAS indicate higher levels of adjustment within a relationship with a partner.
Perceived Stress Scale (PSS) | 6 weeks
  Changes in perceived Stress will be assessed through the Perceived Stress Scale (PSS-14; Cohen, 1994) to examine whether CBT for perinatal anxiety is effective in reducing the extent to which situations in life are perceived as stressful. Items on the PSS-14 are rated on a 5-point scale ranging from 0 (never) to 4 (very often), with total scores ranging from 0-56. Higher scores on the PSS-14 indicate greater levels of perceived stress.
Emotion Regulation Questionnaire (ERQ) | 6 weeks
  Changes in emotion Regulation will be assessed through the Emotion Regulation Questionnaire (ERQ; Gross & John, 20003) and the Difficulties in Emotion Regulation Scale (DERS-II; Gratz & Roemer, 2005) to examine whether CBT for perinatal anxiety has an impact on emotion regulation abilities. Items on the ERQ are rated on a 7-point scale ranging from 1 (strongly disagree) to 7 (strongly agree).The ERQ has two subscales, a Cognitive Reappraisal subscale and an Expressive Suppression subscale. Six items comprise the Cognitive Reappraisal subscale, meaning scores on this subscale range from 6-42. Four items comprise the Expressive Suppression subscale, meaning scores on this subscale range from 4-28.A total score can be obtained by summing the two subscales, meaning the total score range is 10-70. Higher scores indicate greater use of emotion regulation strategies.
WHO Disability Assessment Scale 2.0 (WHODAS) | 6 weeks
  Overall difficulties in functioning will be assessed through the World Health Disability Assessment Schedule 2.0 (WHODAS; WHO, 2010) to examine whether CBT for perinatal anxiety is effective in increasing overall level of functioning. Items on the WHODAS are rated by a clinician on a 5-point scale ranging from 1 (none) to 5 (extreme). Total scores range from 0-60, with greater scores indicating greater disability, or worse overall functioning.
Hamilton Anxiety Scale (HAM-A) | 6 weeks
  The Hamilton Anxiety Scale is an interview format rating scale developed to quantify the severity of anxiety symptomatology and contains a global score (HAM-A; Hamilton, 1956). In the current study, the HAM-A will be used to assess changes in anxiety to examine whether CBT for perinatal anxiety is effective in reducing anxiety symptoms. Items on the HAM-A are scored on a 5-point scale ranging from 0 (not present) to 4 (severe), with a total score range of 0-56. Scores less than 17 indicate mild severity, scores between 18-24 indicate mild to moderate severity and scores between 25-30 indicated moderate to severe anxiety symptoms.
Montgomery-Asberg Depression Scale (MADRS) | 6 weeks
  The Montgomery-Asberg Depression Rating Scale (MADRS; Montgomery & Asberg, 1979) is a measure that requires an interview format assessing depressive symptoms and contains a global severity score. Items on the MADRS are rated on a 6-point scale ranging from 0-6, with total scores ranging from 0-48. Higher total scores indicate greater depressive symptoms.
Difficulties in Emotion Regulation Scale (DERS-II) | 6 weeks
  Changes in emotion regulation will be assessed through the Difficulties in Emotion Regulation Scale (DERS-II; Gratz & Roemer, 2005) and the Emotion Regulation Questionnaire (ERQ, Gross & John, 2003) to examine whether CBT for perinatal anxiety has an impact on emotion regulation abilities. The DERS-II is rated on a 5-point scale ranging from 1 (almost never) to 5 (almost always), with total scores ranging from 39-195. The DERS-II has six factors: Lack of Emotional Awareness (6 items, range 6-30), Lack of Emotional Clarity (5 items, range 5-25), Difficulties Controlling Impulsive Behaviours When Distressed (6 items, range 6-30), Difficulties Engaging in Goal-Directed Behaviour When Distressed (5 items, range, 5-25), Nonacceptance of Negative Emotional Responses (6 items, range 6-30), and Limited Access to Effective ER Strategies (8 items, range 8-40). Total scores are a sum of subscale scores and higher total scores indicate more difficulties with emotion regulation.
Worry Behaviors Inventory (WBI) | 6 weeks
  Changes in anxiety related behaviours (e.g., avoidance and safety behaviours) will be assessed through the Worry Behaviors Inventory (WBI; Mahoney et al., 2016) to examine whether CBT for perinatal anxiety is effective in reducing worry-related behaviours. Items on the WBI are rated on a 5-point scale ranging from 0 (none of the time) to 4 (all of the time), with total scores ranging from 0-40. The WBI has two subscales that measure avoidance (3 items, range 0-12) and safety behaviours (7 items, range 0-28) respectively. Total scores on the WBI are calculated by summing the two subscales. Higher scores indicate greater use of worry related behaviours.
The Female Sexual Function Index (FSFI) | 6 weeks
  Changes in sexual desire, lubrication, orgasm propensity, satisfaction, and pain will be assessed using The Female Sexual Function Index (FSFI; Rosen et al., 2010) to examine whether CBT for perinatal anxiety has an impact on these areas of sexual function. Items one and two on the FSFI are rated on a 5-point scale ranging from 1-5, while items 3-19 are rated on a six-point scale ranging from 0-5. Total scores on the FSFI are obtained by adding the six domain scores together, and range from 2-36. Higher scores on the FSFI indicate lower sexual functioning.
The Sexual Quality of Life - Female (SQoL-F) | 6 weeks
  Changes in sexual quality of life will be assessed using The Sexual Quality of Life - Female (SQoL-F; Symonds et al., 2005) to examine whether CBT for perinatal anxiety has in impact on female sexual dysfunction and women's quality of life. Items on the SQoL-F are scored on a 6-point scale ranging from 1 (completely disagree) to 6 (completely agree). Total scores range from 18-108, with higher scores indicating better female sexual quality of life.
Client Satisfaction Questionnaire (CSQ) | 6 weeks
  Satisfaction of participants receiving CBT for perinatal anxiety will be assessed using the Client Satisfaction Questionnaire (CSQ; Larsen et al., 1979) to examine whether participants are satisfied with the services they have received. Items on the CSQ are rated on a 4-point scale ranging from 1-4. Total scores on the CSQ are a sum ranging from 8-32, with higher scores indicating greater satisfaction with the services received.
Postpartum Bonding Questionnaire (PBQ) | 6 weeks
  Mother-infant bonding will be assessed using the Postpartum Bonding Questionnaire (PBQ; Brockington et al., 2001) to examine whether CBT for perinatal anxiety has an impact on bonding. Items on the PBQ are rated on a 6-point scale ranging from 0 (never) to 5 (always). Total scores on the PBQ range from 0-125. Higher scores on this measure indicate problematic mother-infant bonding.

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl Green, PhD, C.Psych, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- Women's Health Concerns, St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Green SM, Haber E, Frey BN, McCabe RE. Cognitive-behavioral group treatment for perinatal anxiety: a pilot study. Arch Womens Ment Health. 2015 Aug;18(4):631-8. doi: 10.1007/s00737-015-0498-z. Epub 2015 Feb 5. PMID 25652951
- [Derived] Green SM, Donegan E, McCabe RE, Streiner DL, Furtado M, Noble L, Agako A, Frey BN. Cognitive Behavior Therapy for Women With Generalized Anxiety Disorder in the Perinatal Period: Impact on Problematic Behaviors. Behav Ther. 2021 Jul;52(4):907-916. doi: 10.1016/j.beth.2020.11.004. Epub 2020 Nov 20. PMID 34134830